CLINICAL TRIAL: NCT00422682
Title: A Phase 1B, Open-Label, Dose Escalation Study Evaluating the Safety of BSI-201 in Combination With Chemotherapeutic Regimens in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating BSI-201 in Combination With Chemotherapeutic Regimens in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD11484; 20060102 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Tumors
Keywords: Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — iniparib; Topotecan; Temozolomide; Gemcitabine; Carboplatin; Paclitaxel

ARMS (4):
- 1 (Experimental): BSI-201 + topotecan
  Interventions: Drug: bsi-201 + topotecan
- 2 (Experimental): BSI-201 + temozolomide
  Interventions: Drug: bsi-201 + temozolomide
- 3 (Experimental): bsi-201 + gemcitabine
  Interventions: Drug: bsi-201 + gemcitabine
- 4 (Experimental): bsi-201 + carboplatin/paclitaxel
  Interventions: Drug: bsi-201 + carboplatin/paclitaxel

INTERVENTIONS:
Drug: bsi-201 + topotecan — 21 day cycle
  Arms: 1
Drug: bsi-201 + temozolomide — 28 day cycle
  Arms: 2
Drug: bsi-201 + gemcitabine — 28 day cycle
  Arms: 3
Drug: bsi-201 + carboplatin/paclitaxel — 21 day cycle
  Arms: 4

SUMMARY:
The purpose of the study is to assess the safety and establish the maximum tolerated dose (MTD) of the combination of BSI-201 with chemotherapeutic regimens in adult subjects with histologically or cytologically documented advanced solid tumors.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old with a histologically or cytologically documented, advanced solid tumor
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (without granulocyte colony-stimulating factor [G-CSF] support within 2 weeks of study day 1); platelet count ≥ 100.0 x 10^9/L (without transfusion within 2 weeks of study day 1); and hemoglobin ≥ 9.0 g/dL (erythropoietic agents allowed)
* At least a 14-day period from end of last dose of chemotherapy received
* Any prior toxicity from prior chemotherapeutic treatment recovered to ≤ grade 1

Exclusion Criteria:

* Subject enrolled in another investigational device or drug trial, or is receiving other investigational agents
* Hematological malignancies
* Symptomatic or untreated brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and corticosteroids.
* History of seizure disorder
* Myocardial infarction (MI) within 6 months of study day 1, unstable angina, congestive heart failure (CHF) with New York Heart Association (NYHA) > class II, or uncontrolled hypertension
* Concurrent or prior (within 7 days of study day 1) anticoagulation therapy (low dose for port maintenance allowed)
* Specified concomitant medications
* Serum creatinine > 1.5 x upper limit of normal (ULN)
* Elevated liver enzymes (AST/ALT) > 2.5 x ULN, or > 5.0 x ULN if secondary to liver metastases; alkaline phosphatase > 2.5 x ULN or > 5.0 x ULN if secondary to liver or bone metastases; total bilirubin > 1.5 x ULN
* Radiation therapy within 14 days of study day 1
* Antibody therapy for the treatment of an underlying malignancy within 14 days of study day 1
* Concurrent radiation therapy is not permitted throughout the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
safety and efficacy | ongoing
Response rate (CR + PR) | every 2 cycles

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Site, New Haven, Connecticut
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas